CLINICAL TRIAL: NCT06247631
Title: Can the STOP-Bang Questionnaire Predict Obstructive Sleep Apnea and Difficult Mask/Intubation in Patients Scheduled for Thoracic Surgery? Prospective Observational Study
Brief Title: STOP-Bang Questionnaire: A Predictor of Obstructive Sleep Apnea and Difficult Mask/Intubation?
Status: Recruiting | Type: Observational
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Alagoz, Department of anesthesiology and reanimation, Principal Investigator, Specialist Doctor, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Other Study IDs: E-53610172-799-213190410
Record Dates: First submitted 2024-01-22; First posted 2024-02-08 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Difficult Intubation; Airway Disease
Keywords: difficult intubation; difficult mask; Obstructive Sleep Apnea Syndrome; STOP-BANG; thoracic surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: Easy airway: unassisted mask ventilation, ventilation without the need for an airway, achieving oxygen saturation above 90% during mask ventilation, and unassisted intubation with less than three attempts.
  Interventions: Other: STOP BANG
- Difficult airway: Difficult airway: assisted mask ventilation, need for airway during ventilation, oxygen saturation falling below 90% during mask ventilation, assisted intubation, intubation attempt three and above
  Interventions: Other: STOP BANG

INTERVENTIONS:
Other: STOP BANG — The STOP-Bang Questionnaire is intended to give physicians an easy-to-use tool to identify people who might have obstructive sleep apnea (OSA). The questionnaire consists of eight yes-or-no questions based on the major risk factors for OSA. A STOP-Bang score of 2 or less is considered low risk, and a score of 5 or more is high risk for having either moderate or severe OSA. For people who score 3 or 4, doctors may need to perform further assessment to determine how likely they are to have OSA.
  Other Names: STOP-Bang Questionnaire

SUMMARY:
Difficult airway management remains the leading cause of anaesthesia-related morbidity and mortality. Obstructive sleep apnea syndrome (OSAS) is a warning sign of difficult airway management. Polysomnography is the gold standard for diagnosis of this syndrome, but the STOP-BANG questionnaire is the preferred screening test. In this study, we wanted to find an answer to the question How successful is the STOP-BANG questionnaire in screening for obstructive sleep apnea syndrome (OSAS) in predicting OSAS, difficult mask and difficult intubation in patients undergoing thoracic surgery?

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing thoracic surgery
* 18-65 years old
* ASA 1-3

Exclusion Criteria:

* Having a history of obstructive sleep apnea syndrome,
* Having a history of previous head and neck surgery/radiotherapy,
* Patients who did not agree to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-65, ASA 1-3, who will undergo thoracic surgery at the Ankara Atatürk Sanatorium Training and Research Hospital of the University of Health Sciences will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
STOP-BANG questionnaire | 1 month (1 time)
  A STOP-Bang score of 2 or less is considered low risk, and a score of 5 or more is high risk for having either moderate or severe obstructive sleep apnea (OSA). For people who score 3 or 4, doctors may need to perform further assessment to determine how likely they are to have OSA.

CONTACTS AND LOCATIONS:
Overall Officials: Ali ALAGÖZ, professor, Principal Investigator — Ankara Ataturk Sanatorium Training and Research Hospital
Locations (1):
- Ankara Atatürk Sanatorium Training and Research Hospital, Ankara, Keçiören, Turkey (Türkiye)